CLINICAL TRIAL: NCT05382299
Title: A Randomized, Open-label, Phase 3 Study of Sacituzumab Govitecan Versus Treatment of Physician's Choice in Patients With Previously Untreated, Locally Advanced, Inoperable or Metastatic Triple-Negative Breast Cancer Whose Tumors Do Not Express PD-L1 or in Patients Previously Treated With Anti-PD-(L)1 Agents in the Early Setting Whose Tumors Do Express PD-L1
Brief Title: Study of Sacituzumab Govitecan-hziy Versus Treatment of Physician's Choice in Patients With Previously Untreated Locally Advanced Inoperable or Metastatic Triple-Negative Breast Cancer
Acronym: ASCENT-03
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-592-6238; 2021-005743-79 (EudraCT Number); DOH-27082022-7958 (Registry Identifier: South African National Clinical Trials Registry); jRCT2041220122 (Registry Identifier: Japan Registry of Clinical Trials); CTR20234162 (Registry Identifier: China: Drug Clinical Trial Registration and Information Disclosure Platform); 2023-504195-14 (Other: European Medicines Agency)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Triple Negative Breast Cancer; PD-L1 Negative
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab Govitecan-hziy (SG) (Experimental): Participants will receive SG 10 mg/kg on Days 1 and 8 of a 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Treatment of Physician's Choice (TPC) (Active Comparator): Participants will receive TPC determined prior to randomization from 1 of the 3 allowed regimens:
  * Paclitaxel 90 mg/m^2 on Days 1, 8, and 15 of a 28-day cycle
  * Nab-paclitaxel 100 mg/m^2 on Days 1, 8, and 15 of a 28-day cycle
  * Gemcitabine 1000 mg/m^2 + carboplatin area under the curve (AUC) 2 on Days 1 and 8 of a 21-day cycle
  Interventions: Drug: Paclitaxel; Drug: nab-Paclitaxel; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy — Administered intravenously
  Other Names: IMMU-132; Trodelvy™; GS-0132
  Arms: Sacituzumab Govitecan-hziy (SG)
Drug: Paclitaxel — Administered intravenously
  Arms: Treatment of Physician's Choice (TPC)
Drug: nab-Paclitaxel — Administered intravenously
  Other Names: Abraxane®
  Arms: Treatment of Physician's Choice (TPC)
Drug: Gemcitabine — Administered intravenously
  Arms: Treatment of Physician's Choice (TPC)
Drug: Carboplatin — Administered intravenously
  Arms: Treatment of Physician's Choice (TPC)

SUMMARY:
The primary objective of this study is to compare the progression-free survival (PFS) between sacituzumab govitecan-hziy (SG) versus treatment of physician's choice (TPC) in participants with previously untreated, locally advanced, inoperable or metastatic triple-negative breast cancer whose tumors do not express programmed cell death ligand 1 (PD-L1) or in participants previously treated with anti-programmed cell death (ligand or protein) 1 (Anti-PD-(L)1) Agents in the early setting whose tumors do express PD-L1.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals, regardless of race and ethnic group, with previously untreated locally advanced, inoperable or metastatic triple-negative breast cancer (TNBC)

  * Individuals whose tumors are programmed cell death ligand 1 (PD-L1) negative at screening or individuals whose tumors are PD-L1 positive at screening if they have received an anti-PD-(L)1 inhibitor in the (neo) adjuvant setting or if they cannot be treated with a checkpoint inhibitor due to a comorbidity
  * Centrally confirmed TNBC and PD-L1 status on fresh or archival tissue
  * Individuals must have completed treatment for Stage I-III breast cancer, if indicated, and ≥ 6 months must have elapsed (with the exception of endocrine therapy) between completion of treatment with curative intent and first documented local or distant disease recurrence
  * Individuals presenting with de novo metastatic TNBC are eligible
* Measurable disease based on computed tomography (CT) or magnetic resonance imaging (MRI) in accordance with per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. as evaluated locally
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Demonstrates adequate organ function
* Male individuals and female individuals of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception
* Individuals with human immunodeficiency virus (HIV) must be on antiretroviral therapy (ART) and have a well-controlled HIV infection/disease

Key Exclusion Criteria:

* Positive serum pregnancy test or women who are lactating
* Received systemic anticancer treatment within the previous 6 months or radiation therapy within 2 weeks prior to enrollment
* Have not recovered from adverse events (AEs) due to a previously administered agent at the time study entry
* May not be participating in a study with an investigational agent or investigational device within 4 weeks prior to randomization. Individuals participating in observational studies are eligible
* Previously received topoisomerase 1 inhibitors or antibody drug conjugates containing a topoisomerase inhibitor
* Active second malignancy
* Active serious infection requiring antibiotics
* Positive for HIV-1 or 2 with a history of Kaposi sarcoma and/or Multicentric Castleman Disease
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Randomization up to approximately 57 months
  PFS is defined as the time from the date of randomization until the date of objective progressive disease (PD), or death (whichever comes first).

SECONDARY OUTCOMES:
Overall Survival (OS) | Randomization up to approximately 57 months
  OS is defined as the time from the date of randomization until death due to any cause.
Objective Response Rate (ORR) as Assessed by BICR per RECIST Version 1.1 | Randomization up to approximately 57 months
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) that is confirmed at least 4 weeks after initial documentation of response.
Duration of Response (DOR) as Assessed by BICR per RECIST Version 1.1 | Randomization up to approximately 57 months
  DOR is defined as the time from the first documentation of CR or PR to the earlier of the first documentation of definitive PD or death from any cause (whichever comes first).
Time to Response (TTR) as Assessed by BICR per RECIST Version 1.1 | Randomization up to approximately 57 months
  TTR is defined as the time from the date of randomization until the first documentation of CR or PR.
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First dose date up to approximately 57 months plus 30 days
Percentage of Participants Experiencing Clinical Laboratory Abnormalities | First dose date up to approximately 57 months plus 30 days
Change from Baseline in the Physical Functioning Domain as Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, Core Questionnaire, Version 3.0 (EORTC QLQ-C30). | Randomization up to approximately 57 months
  The EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients, it is composed of 30 questions (items) to assess 15 scales; 1 global health status/quality of life (QOL), 5 functional scales (physical, role, cognitive, emotional, and social), and 9 symptom/item scales(fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high/healthy level of function, a high score for the global health status/QOL represents a high QOL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Time to Deterioration (TTD) of Fatigue Scale of the EORTC QLQ-C30 | Randomization up to approximately 57 months
  TTD is defined as the time between the date of randomization and the date of assessment at which a patient experienced a deterioration (≥ 10 points deterioration from baseline in the fatigue scale) or death.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (363):
- United States (130):
  - Arizona Oncology Associates, PC-Hope,1845 W Orange Grove Rd, Tucson, Arizona
  - Arizona Oncology Associates, PC-Hope,2070 W. Rudasill Rd., Tucson, Arizona
  - Arizona Oncology Associates, PC-Hope, Tucson, Arizona
  - Arizona Oncology Associates, PC-Hope,1620 West St. Mary's Road, Tucson, Arizona
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center,201 S. Buena Vista Street, Suite 200, Burbank, California
  - University of California San Diego Moores Cancer, La Jolla, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center,24302 Paseo de Valencia, Suite 200, Laguna Hills, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center,892 Aerovista Place, Suite 240, San Luis Obispo, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center,2020 Santa Monica Blvd, Suite 600, Santa Monica, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center,2336 Santa Monica, Suites 302 and 304, Santa Monica, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center, Santa Monica, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center,1250 La Venta Dr, Suite 100, Westlake Village, California
  - Rocky Mountain Cancer Centers,1700 South Potomac Street, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers,2312 N. Nevada Avenue, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers,6031 E. Woodman Rd., Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers,4700 E. Hale Parkway, Denver, Colorado
  - Rocky Mountain Cancer Centers,11750 West 2nd Place, Lakewood, Colorado
  - Rocky Mountain Cancer Centers,22 West Dry Creek Circle, Littleton, Colorado
  - Rocky Mountain Cancer Centers,10107 Ridge Gate Parkway, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers,2030 Mountain View Ave Ste 210, Longmont, Colorado
  - Rocky Mountain Cancer Centers,3676 Parker Blvd, Pueblo, Colorado
  - Rocky Mountain Cancer Centers,525 W. 15th Street, Pueblo, Colorado
  - Rocky Mountain Cancer Centers,8820 Huron Street, Thornton, Colorado
  - AdventHealth Medical Group, Altamonte Springs, Florida
  - Florida Cancer Specialists - North Region Research Office,750 Orienta Ave, Altamonte Springs, Florida
  - Florida Cancer Specialists,9776 Bonita Beach Road Southeast Suite 201 A, Bonita Springs, Florida
  - Florida Cancer Specialists,3630 Manatee Avenue West, Bradenton, Florida
  - Florida Cancer Specialists,5985 Silver Falls Run, Bradenton, Florida
  - Florida Cancer Specialists - North Region Research Office,403 S. Kings Ave., Brandon, Florida
  - Florida Cancer Specialists,1030 Commerce Creek Blvd, Cape Coral, Florida
  - Florida Cancer Specialists - North Region Research Office,3280 McMullen Booth Road, Clearwater, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists,8981 Colonial Center Drive, Fort Myers, Florida
  - Florida Cancer Specialists,8260 Gladiolus Dr, Fort Myers, Florida
  - Florida Cancer Specialists - North Region Research Office,6420 W. Newberry Road, Gainesville, Florida
  - Florida Cancer Specialists - North Region Research Office,100 Highland Avenue, Largo, Florida
  - Florida Cancer Specialists - North Region Research Office,521 North Lecanto Highway, Lecanto, Florida
  - Florida Cancer Specialists,1100 Goodlette Road, Naples, Florida
  - Florida Cancer Specialists,681 4th Avenue North, Naples, Florida
  - Florida Cancer Specialists - North Region Research Office,4945 SW 49th Place, Ocala, Florida
  - Florida Cancer Specialists - North Region Research Office,2824 Enterprise Rd, Orange City, Florida
  - AdventHealth Medical Group,2501 North Orange Ave, Orlando, Florida
  - Florida Cancer Specialists - North Region Research Office,70 W. Gore Street, Orlando, Florida
  - Florida Cancer Specialists,22395 Edgewater Drive, Port Charlotte, Florida
  - Florida Cancer Specialists,600 North Cattlemen Road, Sarasota, Florida
  - Florida Cancer Specialists,1970 Golf Street, Sarasota, Florida
  - Florida Cancer Specialists - North Region Research Office,7154 Medical Center Drive, Spring Hill, Florida
  - Florida Cancer Specialists - North Region Research Office,1201 Fifth Avenue North, St. Petersburg, Florida
  - Florida Cancer Specialists - North Region Research Office, St. Petersburg, Florida
  - Florida Cancer Specialists - North Region Research Office,3402 West Dr. Martin Luther King Jr. Boulevard, Tampa, Florida
  - Florida Cancer Specialists - North Region Research Office,4100 Waterman Way, Tavares, Florida
  - Florida Cancer Specialists - North Region Research Office,1400 US Highway 441 N, The Villages, Florida
  - Florida Cancer Specialists - North Region Research Office,9320 State Road 54, Trinity, Florida
  - Florida Cancer Specialists,901 South Tamiami Trail, Venice, Florida
  - Florida Cancer Specialists,836 Sunset Lake Blvd, Venice, Florida
  - Florida Cancer Specialists - North Region Research Office,460 N Orlando Ave, Winter Park, Florida
  - Northside Hospital,125 King Avenue, Athens, Georgia
  - Northside Hospital,5670 Peachtree Dunwoody Rd., Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital,308 Deep South Farm Rd, Suite 200, Blairsville, Georgia
  - Northside Hospital,228 Riverstone Dr., Canton, Georgia
  - Northwest Georgia Oncology Northwest Georgia Oncology Centers, PCCenters, PC,157 Clinic Avenue, Carrollton, Georgia
  - Northwest Georgia Oncology Northwest Georgia Oncology Centers, PCCenters, PC,100 Market Place Blvd, Cartersville, Georgia
  - Northside Hospital,1505 Northside Blvd, Suite 4600, Cumming, Georgia
  - Northside Hospital,3855 Pleasant Hill Rd., Suite 480, Duluth, Georgia
  - Northside Hospital,308 Coliseum Dr., Macon, Georgia
  - Northwest Georgia Oncology Northwest Georgia Oncology Centers, PCCenters, PC, Marietta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,1 Kish Hospital Drive, DeKalb, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,10 Health Services Drive, DeKalb, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,300 Randall Road, Geneva, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,304 Randall Road, Geneva, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,1000 N. Westmoreland Road, Lake Forest, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,4405 Weaver Parkway, Warrenville, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,4455 Weaver Parkway, Warrenville, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,25 N Winfield Road, Winfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Norton Cancer Institute - Saint Matthews,234 E. Gray Strret, Louisville, Kentucky
  - Norton Cancer Institute - Saint Matthews,676 S. Floyd Street, Louisville, Kentucky
  - Norton Cancer Institute - Saint Matthews, Louisville, Kentucky
  - Norton Cancer Institute - Saint Matthews,4955 Norton Healthcare Blvd, Louisville, Kentucky
  - Cancer Institute Ascension Saint Agnes, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - The West Clinic, PLLC dba West Cancer Center,7668 Airways Blvd, Southaven, Mississippi
  - New York Cancer & Blood Specialists - Port Jeffers,72 East Main St., Babylon, New York
  - New York Cancer & Blood Specialists - Port Jeffers,1 Delaware Dr., New Hyde Park, New York
  - New York Cancer & Blood Specialists - Port Jeffers,365 East Main St., Patchogue, New York
  - New York Cancer & Blood Specialists - Port Jeffers,1500 Rte, 112, Building 4, Port Jefferson, New York
  - New York Cancer & Blood Specialists - Port Jeffers,49 Rte. 347, Newconset Hwy, Port Jefferson Station, New York
  - New York Cancer & Blood Specialists - Port Jeffers, Port Jefferson Station, New York
  - New York Cancer & Blood Specialists - Port Jeffers,750 Old County Rd. Suite 4, Riverhead, New York
  - New York Cancer & Blood Specialists - Port Jeffers,12 East 86th St, Suite 4, The Bronx, New York
  - New York Cancer & Blood Specialists - Port Jeffers,2330 Eastchester Road, Suite 360, The Bronx, New York
  - Novant Health Cancer Institute - Forsyth,125 Queens Road, Suite 650, Charlotte, North Carolina
  - Novant Health Cancer Institute - Forsyth,2131 S. 17th Street, Wilmington, North Carolina
  - Novant Health Cancer Institute - Forsyth, Winston-Salem, North Carolina
  - Magee-Womens Hospital of UPMC,2500 West 12th Street, Erie, Pennsylvania
  - Magee-Womens Hospital of UPMC,201 State Street, 6 Main, Erie, Pennsylvania
  - Magee-Womens Hospital of UPMC,4300 Londonberry Road, Harrisburg, Pennsylvania
  - Magee-Womens Hospital of UPMC,2035 Technology Parkway, Mechanicsburg, Pennsylvania
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital of UPMC,5115 Centre Avenue, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital of UPMC,1703 Innovation Drive, York, Pennsylvania
  - Tennessee Oncology, PLLC,103 Natchez Park Drive, Dickson, Tennessee
  - Tennessee Oncology, PLLC,4488 Carothers Parkway, Franklin, Tennessee
  - Tennessee Oncology, PLLC,225 Big Station Camp Blvd, Gallatin, Tennessee
  - The West Clinic, PLLC dba West Cancer Center, Germantown, Tennessee
  - Tennessee Oncology, PLLC,353 New Shackle Island Road, Hendersonville, Tennessee
  - Tennessee Oncology, PLLC,5653 First Blvd., Hermitage, Tennessee
  - Tennessee Oncology, PLLC,103 Physicians Way, Lebanon, Tennessee
  - Tennessee Oncology, PLLC,1840 Medical Center Parkway, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC,2004 Hayes Street, Nashville, Tennessee
  - Tennessee Oncology, PLLC,SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Tennessee Oncology, PLLC,4220 Harding Rd, Nashville, Tennessee
  - Tennessee Oncology, PLLC,3443 Dickerson Road, Nashville, Tennessee
  - Tennessee Oncology, PLLC,397 Wallace Road, Nashville, Tennessee
  - Tennessee Oncology, PLLC,120 Frank Martin Road, Shelbyville, Tennessee
  - Tennessee Oncology, PLLC,300 Stonecrest Blvd, Smyrna, Tennessee
  - Texas Oncology PA,901 West 38th Street, Austin, Texas
  - Texas Oncology PA, Austin, Texas
  - Texas Oncology PA,4101 James Casey, Suite 100, Austin, Texas
  - Virginia Oncology Associates,744 N. Battlefield Blvd, Chesapeake, Virginia
  - Virginia Oncology Associates,1051 Loftis Blvd Suite 100, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Oncology Associates,1950 Glenn Mitchell Drive, Virginia Beach, Virginia
- Argentina (6):
  - Hospital Británico de Buenos Aires, Buenos Aires
  - Instituto de Oncologia Angel H.Roffo, CABA
  - Fundacion CORI para la Investigacion y Prevencion del Cancer, Capital
  - Instituto de Oncología de Rosario, Rosario
  - Centro para la Atencion Integral del Paciente Oncologico Centro Médico C.A.I.P.O, San Miguel de Tucumán
  - Clinica Viedma, Viedma
- Australia (7):
  - Saint George Hospital - Australia, Kogarah, New South Wales
  - Mater Misericordiae Limited and Mater Research Limited, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Cancer Research SA (CRSA), Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Austin Hospital, Melbourne, Victoria
  - Breast Cancer Research Center - Western Australia, Nedlands, Western Australia
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz
- Belgium (7):
  - Algemeen Ziekenhuis Klina, Brasschaat
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Grand Hopital de Charleroi - Notre Dame, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire Université Cathol, Namur
- Brazil (14):
  - Hospital Araújo Jorge - Associação de Combate ao Câncer em Goiás - ACCG, Goiânia
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí
  - Catarina Pesquisa Clínica, Itajaí
  - Hospital Moinhos de Vento, Porto Alegre
  - Hospital de Clinicas de Porto Alegre - HCPA, Porto Alegre
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Instituto Nacional de Câncer - INCA - HCIII, Rio de Janeiro
  - Núcleo de Oncologia da Bahia, Salvador
  - CEPHO - Centro de Estudos e PesquisaS de Hematologia e Oncologia, Santo André
  - Real e Portuguesa de Beneficéncia - Hospital Beneficéncia Portuguesa (BP) - Unidade Paulista, São Paulo
  - Clinica de Pesquisas e Centro de Estudos em Oncolo, São Paulo
  - Fundação Pio XII - Hospital de Amor de Barretos, São Paulo
  - Hospital Amaral Carvalho, São Paulo
  - Nucleo de Pesquisa Clinica da Rede Sao Camilo, São Paulo
- Canada (9):
  - Cross Cancer Institute, Edmonton
  - QEII Health Sciences Centre, Halifax
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchener
  - London Health Sciences Centre, London
  - Jewish General Hospital Department of Medical Oncology, Montreal
  - McGill University Health Centre, Montreal
  - Ottawa Hospital - General Campus, Ottawa
  - Sunnybrook Research Institute, Toronto
  - Mount Sinai Hospital, Toronto
- Chile (5):
  - Oncovida - Santiago, Providencia
  - Clínica Alemana, Santiago
  - Clínica IRAM, Santiago
  - Centro de Oncología de Precisión, Santiago Region
  - James Lind Centro de Investigacion del Cancer, Temuco
- China (28):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - The First Medical Center of Chinese PLA General Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Chongqing University Cancer Hospital, Chongqing
  - Deyang People's Hospital, Deyang
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Cancer Hospital, Hefei
  - The Second Hospital of Anhui Medical University, Hefei
  - The Second Hospital of Jilin University, Jilin Sheng
  - The Second Hospital of Shandong University, Jinan
  - Shandong Cancer Hospital, Jinan
  - Nanchang People's hospital, Nanchang
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Tianjin Medical University Cancer Institute& Hospital, Tianjin
  - Weihai Municipal Hospital, Weihai
  - Hubei Cancer Hospital, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Zhejiang
- Czechia (6):
  - Masarykuv onkologicky ustav, klinika komplexni onkologickie pece, Brno
  - Fakultni nemocnice Hradec Kravlove, Klinika onkologie a radioterapie, Hradec Králové
  - Fakultní Thomayerova nemocnice, Hradec Králové
  - Fakultni nemocnice Olomouc, Onkologicka klinika, Olomouc
  - Fakultni nemocnice Karlovske Vinohrady, Radioterapeuticka a onkologicka klinika, Prague
  - Vseobecna Fakultni Nemocnice v Praze, Prague
- France (12):
  - Sainte Catherine Institut du Cancer Avignon Provence, Avignon
  - Centre Hospitalier Régional et Universitaire de Be, Besançon
  - Hôpital Morvan, Institut de cancérologie, Brest
  - Centre francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Cancérologie du Grand Montpellier, Montpellier
  - Hôpital Privé du Confluent, Nantes
  - Hospices Civils de Lyon Hôpital Lyon Sud, Pierre-Bénite
  - Centre Armoricain de Radiothérapie, dImagerie Méd, Plérin
  - Centre Eugène Marquis, Rennes
  - Institut Claudius Regaud - IUCT-O, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (9):
  - Helios Klinikum Berlin-Buch, Berlin
  - Gynakologisches Zentrum Bonn, Schwerpunkt Gyn. Onkologie,, Bonn
  - Klinik Frauenheilkunde, Uniklinik ClO, Studienzentrale, Cologne
  - Kliniken Essen-Mitte - Evangelische Huyssens-Stift Breast Unit, Essen
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Nationales Centrum für Tumorerkrankungen - Heidelb, Heidelberg
  - Universitätsklinikum Schleswig-Holstein Institut fur Klinische Chermie, Lübeck
  - Universitatsklinikum Mannheim GmBH, Frauenklinik, Mannheim
  - Universitätsklinikum Tübingen, Tübingen
- Hong Kong (3):
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - Queen Mary Hospital, Pok Fu Lam
- Hungary (3):
  - Uzsoki Utcai Kornaz, Onkoradiologiai Osztaly, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Petz Aladar Egyetemi Oktaté Kérhaz - Osztaly, Győr
- Israel (7):
  - Rambam Health Care Campus, Haifa
  - Hadassah - Hebrew University Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Sheba Medical Center Hospital - Tel Hashomer, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (15):
  - IRCCS Istituto Tumori "G.Paolo II", Bari
  - SSD Oncologia Medica Addarii-Zamagni, IRCSS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant'Orsola, Bologna
  - UO Oncologia, ASST degli Spedali Civili di Brescia, Brescia
  - IRCSS Ospedale Policlinico San Martino, Genova GE
  - S.C. Oncologia medica, ASST di Lecco, Lecco
  - Presidio Ospedaliero di Lucca, Lucca
  - Ospedale Generale Provinciale - Macerata, Macerata
  - Istituto Europeo di Oncologia, Milan
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
  - Azienda Socio Sanitaria Territoriale, Monza
  - Oncologia Medica Senologica Sperimentale - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Azienda Ospedaliero-Universitaria Maggiore della C, Novara
  - Istituto Oncologico Veneto - IRCCS, Padua
  - AOU Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario Agostino Geme, Rome
- Japan (20):
  - Aichi Cancer Center Hospital, Aichi
  - Juntendo University Hospital, Bunkyō City
  - Chiba Cancer Center, Chūōku
  - Shikoku Cancer Center, Ehime
  - Hakuaikai Sagara Hospital, Kagoshima
  - National Cancer Center Hospital East, Kashiwa
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Kumamoto University Hospital, Kumamoto
  - Kure Medical Center And Chugoku Cancer Center, Kure
  - National Hospital Organization Kyushu Cancer Center, Minamiku
  - Nagoya University Hospital, Nagoya
  - Hiroshima City Hiroshima Citizens Hospital, Nakaku
  - Okayama University Hospital, Okayama
  - Kyoto University Hospital, Sakyo-ku
  - Hokkaido Cancer Center, Sapporo
  - Shizuoka Cancer Center, Shizuoka
  - Shizuoka General Hospital, Shizuoka
  - Osaka University Hospital, Suita
  - Showa University Hospital, Tokyo
  - Kanagawa Cancer Center, Yokohama
- Malaysia (7):
  - Hospital Pulau Pinang, George Town
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre (UMMC), Kuala Lumpur
  - Institut Kanser Negara, Putrajaya
  - Sarawak General Hospital, Sarawak
- Mexico (10):
  - Icaro Investigaciones en Medicina, Chihuahua City
  - Sinacor - Centro para el Desarrollo de la Medicina, Culiacán
  - Panamerican Clinical Research Mexico - Guadalajara, Guadalajara
  - Cryptex Investigación Clínica, Mexico City
  - Medical Care and Research S.A. de C.V., Mérida
  - Fucam A.C., México
  - Avix Investigacion Clinica S.C., Monterrey
  - Oncológico Potosino, San Luis Potosí City
  - FAICIC Clínical Research, Veracruz
  - iBiomed - Investigacion Biomedica para el Desarrol, Zapopan
- Netherlands (5):
  - Amphia Ziekenhuis - Breda Langendijk, Breda
  - Universitair Medisch Centrum Groningen, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej, Gliwice
  - SP ZOZ Opolskie Centrum Onkologii im. prof. Tadeusza Koszarowskiego, Opole
  - Mazowiecki Szpital Wojewódzki im. w. Jana Pawa II, Siedlce
  - Narodowy Instytut Onkologii im.Marii Marii Sklodowskiej, Warsaw
- Romania (4):
  - Spitalul Clinic Filantropia, Bucharest
  - SC Medisprof SRL, Cluj-Napoca
  - Institutal Oncologic, Prof. Dr Ion Chiricuta, Cluj-Napoca
  - Centrul De Oncologie Sf Nectarie, Craiova
- Slovakia (3):
  - Onkologicky Ustav Sv. Alzbety, Bratislava
  - Národný onkologický ústav, Bratislava
  - Nemocnica Partizánske, Partizánske
- South Africa (3):
  - Hopelands Cancer Centre, Hilton
  - Wits Clinical Research, Johannesburg
  - The Medical Oncology Centre of Rosebank, Johannesburg
- South Korea (8):
  - National Cancer Center, Goyang-si Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Spain (13):
  - Hospital Teresa Herrera - Materno Infantil, A Coruña
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Maranon, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Unviersitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
- Kantonsspital St.Gallen, Sankt Gallen, Switzerland
- Taiwan (7):
  - Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital, Lioying, Tainan
  - National Taiwan University Hospital, Taipei
  - MacKay Medical Foundation The Presbyterian Church in Taiwan MacKay Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- Turkey (Türkiye) (11):
  - Baskent Uni. Dr Turgut Noyan Uyg. ve Aras. Merkezi, Adana
  - Memorial Ankara Hastanesi, Ankara
  - Ankara Il Saglik Mudurlugu SBU Gulhane Egitim Ve A, Ankara
  - Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi, Ankara
  - Hacettepe Üniversitesi Hastanesi, Ankara
  - Trakya Universitesi Tip Fakultesi Hastanesi, Edirne
  - Istanbul Il Saglik Mudurlugu Goztepe Prof. Dr. Sul, Istanbul
  - Medipol Mega Universite Hastanesi, Istanbul
  - Ege Universitesi Hastanesi, Izmir
  - Medicana International Izmir Hastanesi, Izmir
  - Acibadem Maslak Hastanesi, Sarıyer
- United Kingdom (3):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Barts Health NHS Trust, London
  - University College London Hospitals NHS Foundation, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cortes J, Punie K, Barrios C, Hurvitz SA, Schneeweiss A, Sohn J, Tokunaga E, Brufsky A, Park YH, Xu B, Hegg R, Oliveira M, Fabi A, Vaksman N, Valdez T, Zhang X, Lai C, Tolaney SM; ASCENT-03 Clinical Trial Investigators. Sacituzumab Govitecan in Untreated, Advanced Triple-Negative Breast Cancer. N Engl J Med. 2025 Nov 13;393(19):1912-1925. doi: 10.1056/NEJMoa2511734. Epub 2025 Oct 19. PMID 41124233
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-592-6238